CLINICAL TRIAL: NCT01874236
Title: VaReFi Validity and Reliability of Diagnostic Findings of SI Joint Blocking
Brief Title: Validity and Reliability of Diagnostic Findings of SI Joint Blocking
Acronym: VaReFi
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Data could not be interpreted. Re-design efforts failed.
Sponsor: SI-BONE, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 300164
Record Dates: First submitted 2013-05-30; First posted 2013-06-10 (Estimated); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: SI Joint Pain
Keywords: SI joint pain, SI joint dysfunction, degenerative sacroiliitis, sacroiliac joint disruption
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1st sequence (Active Comparator): Blinded 3 blocks (2 bupivacaine, 1 sham block)
  Interventions: Drug: 0.75% bupivacaine
- 2nd sequence (Active Comparator): Blinded 3 blocks (2 bupivacaine, 1 sham block)
  Interventions: Drug: .75% bupivacaine
- 3rd sequence (Active Comparator): Blinded 3 blocks (2 bupivacaine, 1 sham block)
  Interventions: Drug: .75% bupivacaine

INTERVENTIONS:
Drug: 0.75% bupivacaine — Week 1: SI joint injection with .75% bupivacaine Week 2: SI joint injection with .75% bupivacaine Week 3: SI joint sham block
  Other Names: Blinded 3 blocks (2 bupivacaine, 1 sham block)
  Arms: 1st sequence
Drug: .75% bupivacaine — Week 1: SI join sham block Week 2: SI joint injection with .75% bupivacaine Week 3: SI joint injection with .75% bupivacaine
  Other Names: Blinded 3 blocks (2 bupivacaine, 1 sham block)
  Arms: 2nd sequence
Drug: .75% bupivacaine — Week 1: SI join injection with .75% bupivacaine Week 2: SI join sham block Week 3: SI joint injection with .75% bupivacaine
  Other Names: Blinded 3 blocks (2 .75% bupivacaine, 1 sham block)
  Arms: 3rd sequence

SUMMARY:
The purpose of the trial is to confirm the validity and reliability of diagnostic SI joint blocks.

DETAILED DESCRIPTION:
Subjects with suspected SI joint pain will undergo 3 SI joint blocks, 2 with local anesthetic and 1 sham block.

The sequence of blocks is randomly assigned. This study examines both the test-retest reliability of response to diagnostic sacroiliac (SI) joint injection and the specificity of response to local anesthetic or sham block. The goal of the study is to validate the use of diagnostic SI joint block.

Subjects with pain suspected to be generated by one SI joint will undergo three diagnostic SI joint blocks each separated by one week. Two blocks will be with local anesthetic (LA) and one will be a sham block (SB). Both the Coordinator (collecting pain assessments) and subject will be blinded to the sequence of blocks (LA or SB each time). The sequence of blocks will be randomly assigned for each subject on study. The subject's participation in the study is complete after 6-month post-procedure assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21-75 at time of screening.
2. Patient has buttocks, groin and/or leg pain suspected to be from one SI joint (left or right).
3. Patient has positive Fortin finger test*.
4. Patient has a current average SI joint pain rating of at least 5 on 0-10 numerical rating scale**.
5. Patient has at least 3 positive physical SI joint examination findings in the targeted SI joint.
6. Investigator believes that diagnostic SI joint block is indicated now, and that no other (hip/back, etc.) diagnostic test is required at this time.
7. Patient has signed study-specific informed consent form.
8. Patient has the necessary mental capacity to participate and is physically able to comply with study protocol requirements (including avoiding taking pain medication 8 hours prior to and 4 hours after each scheduled block).

Exclusion Criteria:

1. Patient has history of any surgical procedure of the targeted SI joint (except for prior RF ablation of the SI joint).
2. Patient has suspected bilateral SIJ pain and bilateral injections are indicated.
3. Patient has history of chronic pain syndrome (e.g., fibromyalgia).
4. Patient has any medical or other condition that would interfere with study participation or data validity.
5. Patient is currently pregnant.
6. Patient has known allergy to contrast used or local anesthetic used (bupivacaine).
7. Patient has had one or more steroid SI joint injection(s) of the targeted side in the last 3 months.
8. Patient is a prisoner or a ward of the state.
9. Patient is participating in another investigational study related to back or SI joint pain (Exclude if participating in trials other than the SIFI study (NCT01640353) or the INSITE Study (NCT01681004). Subjects on these two SI-BONE sponsored trials may be eligible for VaReFi.)
10. Patient is known or suspected drug or alcohol abuser.
11. Patient has known or suspected psychiatric disease (e.g., schizophrenia, major depression, personality disorders) that could interfere with study participation .
12. Patient is unable to isolate suspected SI joint pain to the SI joint but rather has generalized pain.
13. Patient has known or suspected alternative cause for pain at/near SI joint (e.g., lumbar disc degeneration, lumbar facet arthropathy, hip osteoarthritis or labral tear)

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2013-04-22 (Actual); Primary Completion 2014-09-30 (Actual); Study Completion 2014-09-30 (Actual)

PRIMARY OUTCOMES:
Numeric Rating Scale | Baseline, 30 minutes and 60 minutes, 2 and 4 hours post injection (x 3 injections, each 1 week apart), and 1 month post 3rd injection visit (7 weeks post 1st injection).
  Change in SI joint pain from prior to injection to 30 minutes, 60 minutes, 2 hours, 4 hours after injection. Changes compared over 3 injections, where type of block is blinded.
  Is response to bupivacaine different than response to sham block Is response to bupivacaine during second injection similar to that during first injection?

SECONDARY OUTCOMES:
Subgroup analysis by diagnosis at 1 month post 3rd block (7 weeks post 1st injection) and 6 month post 3rd injection visit ( 27 weeks post 1st injection). | 7 weeks after 1st block & and 27 weeks after 1st block
  Look at responses in patients who have been diagnosed with an SI joint condition vs. patients who have no SI joint condition diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Calodney, MD, Principal Investigator — Texas Spine and Joint Hospital
Locations (7):
- United States (7):
  - Orthopedic Center of Southern Illinois, Mount Vernon, Illinois
  - Bluegrass Orthopaedics and Hand Care Research, LLC, Lexington, Kentucky
  - Cleveland Clinic, Cleveland, Ohio
  - Penn State College Of Medicine, Hershey, Pennsylvania
  - Precision Spine Care, Tyler, Texas
  - Physicians' Research Options, LLC, Sandy City, Utah
  - Virginia iSpine Research Institute, Inc, Richmond, Virginia